CLINICAL TRIAL: NCT01758705
Title: Observational Study; Clinical Effectiveness and Impact on Patient Reported Outcomes in Venezuelan Patients With Psoriasis After 16 Weeks of ADA Therapy
Brief Title: Post Marketing Observational Study on Venezuelan Patients With Psoriasis
Status: Withdrawn | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P13-709
Record Dates: First submitted 2012-12-26; First posted 2013-01-01 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Moderate to Severe Chronic Plaque Psoriasis
Keywords: Psoriasis; Related to Health Quality of Life; Patient Reported Outcomes; Venezuelan Patients
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Cohort 1

SUMMARY:
The aim of this study is to obtain Venezuelan data of clinical effectiveness, impact in the HRQoL, work productivity and activity impairment in patients with psoriasis using adalimumab.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with moderate to severe chronic plaque psoriasis, with or without psoriatic arthritis, who have the indication for adalimumab because they need systemic therapy or because they have had failure to phototherapy, or to other systemic or topical treatments
* Subjects that are not receiving biologic therapy in the last 12 weeks or classical therapy in the past 4 weeks and/or phototherapy in the last 2 weeks. Topical therapy will be allowed, to a constant dose and will not be used within 24 hours prior to the visit
* Patients under previous treatment with any experimental drug will have a minimum washout period of five half-lives
* Subjects must be capable to understand and willing to give a written informed consent form to release information and to comply with the requirements of the study protocol

Exclusion Criteria:

* Subjects should not be enrolled if they cannot be treated in accordance with the local product label approved in Venezuela
* Subjects enrolled into another study or under treatment with an investigational product
* History of viral hepatitis B infection or HIV
* History of neurologic symptoms suggestive of central nervous system demyelinating disease
* History of cancer or lymphoproliferative disease (other than successfully treated non-melanoma skin cancer or localized carcinoma in situ of the cervix)
* Active TB infection before initiating adalimumab treatment or latent TB infection not able to complete prophylactic treatment
* Pregnant or lactating female. Pregnancy will be tested before entering the study in fertile women. Women in fertile age must be advised by the physician, to use a clinically accepted contraceptive method (contraceptive pills, IUDs, barrier devices as condoms or abstinence)
* History of congestive heart failure (CHF)
* Any another condition that according to the criteria of the participating investigator represents an obstacle for study conduction and / or subjects to an unacceptable risks
* Subjects with active infection including chronic or localized infections until infections are controlled
* History of sensitive to latex or other component of the syringe
* Subjects who requires concomitant phototherapy and systemic therapy during adalimumab therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects male or female with moderate to severe chronic plaque psoriasis with or without psoriatic arthritis. Patients with history of psoriatic arthritis or articular symptoms must be evaluated by a Rheumatologist.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in PASI 75 (Psoriasis Area and Severity Index score) Response Rate | From Week 0 to Week 16
Change in Percentage of patients with clinical difference in DLQI (Dermatology Life Quality Index) score | From Week 0 to Week 16
  Clinical difference is defined by a minimal important difference (MID) in DLQI score between 2.3-5 at 16 weeks

SECONDARY OUTCOMES:
Mean change of PASI score | From week 0 to week 16
Mean change of DLQI score | From week 0 to week 16
Changes in Psoriatic Arthritis Response Criteria (PsARC) score | From week 0 to week 16
Mean change of Hospital Anxiety and Depression Score (HADS) | From week 0 to week 16
Mean change en Work Productivity and Activity Impairment (WPAI)-Psoriasis score | From week 0 to week 16
Percentage of subjects with Serious Adverse Events (SAEs) | Up to week 16
  Occurrence of SAEs including tuberculosis, other opportunistic infections and cancer
Discontinuation of adalimumab for any reason. | Up to week 16

CONTACTS AND LOCATIONS:
Overall Officials: Natali Serra-Bonett, MD, Study Chair — Abbott